CLINICAL TRIAL: NCT06604871
Title: Safety Evaluation of the MiniMed™ 780G System Used in Combination With the DS5 CGM in Children 2-6 Years of Age
Brief Title: Safety Evaluation of MiniMed™ 780G System With DS5 CGM in Children
Acronym: SUCCEED2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP344
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MiniMed™ 780G system with DS5 (Experimental): Subjects 2-6 years old with type 1 diabetes wearing the MiniMed™ 780G insulin pump in combination with the DS5 CGM.
  Interventions: Device: Insulin Pump with Continuous Glucose Monitoring

INTERVENTIONS:
Device: Insulin Pump with Continuous Glucose Monitoring — MiniMed™ 780G insulin pump in combination with the DS5 CGM

SUMMARY:
The purpose of this study is to evaluate the safety of the MiniMed 780G insulin pump used in combination with the DS5 CGM in type 1 pediatric subjects (2-6 years of age) in a home setting.

DETAILED DESCRIPTION:
This study is a multi-center, single arm study in insulin-requiring pediatric subjects with type 1 diabetes on the MiniMed 780G system using DS5. The run-in period and study period, together, will be approximately 130 days long.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2-6 years at time of screening.
2. Has a clinical diagnosis of type 1 diabetes for 3 months or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
3. Parent(s)/guardian(s) is/are literate and able to read the language offered in the pump or pump materials.
4. Subject or parent(s)/guardian(s) is/are willing to provide informed consent for participation.
5. Is willing to perform fingerstick blood glucose measurements as needed.
6. Is willing to wear the system continuously throughout the study.
7. Must have a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 6 units on average.
8. Has a Glycosylated hemoglobin (HbA1c) less than 10% (as processed by Central Lab) at time of screening visit.

   Note: All HbA1c blood specimens will be collected via fingerstick and sent to and tested by a National Glycohemoglobin Standardization Program (NGSP) certified Central Laboratory. HbA1c testing must follow NGSP standards.
9. Is willing to upload data from the study pump, must have Internet access, and a computer system, or compatible smartphone that meets the requirements for uploading the study pump.
10. Is willing to take one of the following insulins and can financially support the use of insulin preparations as required by the study per manufacturers labeling:

    1. Humalog (insulin lispro injection)
    2. Authorized generic insulin lispro
    3. NovoLog (insulin aspart injection)
    4. Authorized generic insulin aspart
    5. Admelog (insulin lispro injection) - for subjects aged 3 years and older only
11. Has 1 month or more of CGM experience at time of screening.
12. If subject has been diagnosed with hyperthyroidism or hypothyroidism, he/she must have a TSH within 3 months prior to screening or at time of screening.

Exclusion Criteria:

1. Has a history of 1 or more episodes of severe hypoglycemia during the 3 months prior to screening.
2. Has been hospitalized or has visited the emergency room (ER) in the 3 months prior to screening resulting with a primary diagnosis of uncontrolled diabetes.
3. Has had DKA in the last 3 months prior to screening visit.
4. Will not tolerate tape adhesive in the area of sensor placement as assessed by a qualified individual.
5. Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
6. Has diagnosis of adrenal insufficiency.
7. Has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.
8. Is using hydroxyurea at time of screening or plans to use it during the study.
9. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks.
10. Is using pramlintide (Symlin), DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of screening.
11. Parent(s)/guardian(s) has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator.
12. Has elective surgery planned that requires general anesthesia during the course of the study.
13. Has sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening.
14. Plans to receive red blood cell transfusion or erythropoietin over the course of study participation.
15. Is diagnosed with current eating disorder such as anorexia or bulimia.
16. History of chronic renal disease or currently on hemodialysis
17. Has hemophilia or any other bleeding disorder.
18. Has celiac disease that is not adequately treated as determined by the investigator.
19. Has a cardiovascular condition which the investigator determines must exclude the subject.
20. Has hyperthyroidism or hypothyroidism that is not adequately treated as determined by the investigator.
21. Is an immediate family member of a Medtronic Diabetes employee.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint - Percent of Time in Range (TIR 70-180 mg/dL) | Last 6-7 weeks of study period.
  Percent of Time in Range (TIR 70-180 mg/dL). Descriptive only.
Primary Safety Endpoints - Incidence of Adverse Events | Through study completion, approximately 18 months.
  The safety data associated with diabetes management will be summarized:
  * Serious Adverse Events (SAE)
  * Serious Adverse Device Effects (SADE)
  * Unanticipated Adverse Device Effects
  * Incidence of Severe Hypoglycemia
  * Incidence of Severe Hyperglycemia
  * Incidence of DKA
  The details of all AEs will also be presented under Reported Adverse Events in ClinicalTrials.gov.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Stanford University, Palo Alto, California
  - UCSF The Madison Clinic for Pediatric Diabetes, San Francisco, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Nemours Childrens Specialty Care, Jacksonville, Florida
  - USF Diabetes and Endocrinology Center, Tampa, Florida
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Texas Childrens Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No